CLINICAL TRIAL: NCT01836263
Title: Prevention and Treatment of Digital Ulcers in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: marco matucci cerinic (Other)
Collaborators: European Union (Other); University of Giessen (Other); University of Zurich (Other); University of Paris 5 - Rene Descartes (Other); University of Campania Luigi Vanvitelli (Other); University of Basel (Other); University College, London (Other); Charite University, Berlin, Germany (Other); University of Pecs (Other); University of Leeds (Other); Schoen Klinik Hamburg Eilbek (Other)
Responsible Party: Sponsor-Investigator, marco matucci cerinic, Prof. Marco Matucci-Cerinic, University of Florence
Organization: University of Florence (Other)
Other Study IDs: HEALTH-F5-2012-305495-OT1
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Sclerosis; Ulcer
MeSH Terms: conditions — Scleroderma, Systemic; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prevention arm: CCB & i.v. iloprost: prevention arm: patients receiving a combination of calcium channel blockers (CCB) and concomitant i.v. iloprost (i.v. iloprost at least in the last three months)
- Prevention arm: bosentan & sildenafil: prevention arm: patients receiving a combination of the endothelin receptor antagonist bosentan and the Phosphodiesterase-5 inhibitor sildenafil
- Healing arm: CCB & i.v. iloprost: healing arm: patients receiving a combination of calcium channel blockers (CCB) and concomitant i.v. iloprost (i.v. iloprost at least in the last three months)
- Healing arm: bosentan & sildenafil: healing arm: patients receiving a combination of the endothelin receptor antagonist bosentan and the Phosphodiesterase-5 inhibitor sildenafil

SUMMARY:
Systemic sclerosis is an orphan, multiorgan disease affecting the connective tissue of the skin and several internal organs.

Digital ulcers are frequent and have a major impact on the quality of life in patients with systemic sclerosis. The etiology of digital ulcers is complex and multifactorial and the principal mechanisms underlying the digital ulcers formation are ischemic, mechanic and inflammatory, alone or in combination, on the basis of the systemic sclerosis vasculopathy. Consequently, there are at least three types of DU: (i) those localized at the tips of the fingers and toes, mainly resulting from an ischemic process, (ii) those localized on the dorsal aspect of the fingers where the skin retraction due to fibrosis over bony prominences seems to be the main cause, and (iii) those evolving on a pitting scar or subcutaneous calcinosis due to a combined irritative-inflammatory mechanism. An early therapy to prevent or rapidly heal digital ulcers is today considered a mandatory approach to maintain quality of life and spare the enormous costs due to conventional digital ulcer management.

This observational trial is part of the collaborative project "DeSScipher", one out of five observational trials to decipher the optimal management of systemic sclerosis.

Aim of this observational trial is:

1. To identify the best treatment combination for prevention of digital ulcers in patients with fulfilment of the new ACR/EULAR SSc criteria or the preliminary VEDOSS criteria for very early diagnosis of systemic sclerosis
2. To identify the best treatment associated with improved healing of digital ulcers in patients with fulfilment of the new ACR/EULAR SSc criteria

Thus, the observational trial consist of a prevention arm and a healing arm.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile and adult patients with diagnosis of systemic sclerosis according to the ACR/EULAR SSc criteria or the PRES/ACR/EULAR juvenile SSc criteria for enrollment into the prevention and healing arm
* Patients with fulfilment of the preliminary criteria for very eary diagnosis of systemic sclerosis (VEDOSS criteria) for enrollment into the prevention arm

Patients with active digital ulcers will be allocated into the healing arm. Patients without previous or history of digital ulcers (but currently without active digital ulcers) will be allocated into the prevention arm.

Definition of digital ulcers (DU): DU are 1) loss of tissue, 2) DU derived from digital pitting scars and 3) DU derived from calcinosis.

IN THIS STUDY WE CONSIDER ONLY DU (1) LOSS OF TISSUE. THE OTHER DU (2) and DU (3) ARE REGISTERED IN THE DATA BASE IF THEY ARE PRESENT, BUT ARE EXCLUDED FROM EVALUATION.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are adult and juvenile systemic sclerosis patients from the EUSTAR cohort (MEDSonline database), the VEDOSS cohort and the jSScWG cohort
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Prevention arm: Number of new digital ulcers | 24 months
Healing arm: Time to healing of manifest digital ulcers | 24 months

SECONDARY OUTCOMES:
Prevention arm: Time to development of new digital ulcers | 24 months
Healing arm: Number of healed digital ulcers | 24 months

OTHER OUTCOMES:
Prevention arm: novel composite digital ulcer prediction score | 24 months
  Prevention: A novel composite digital ulcers prediction score which will be tested against the already proposed capillaroscopic prediction score CSURI
Healing arm: novel composite outcome score for the assessment of worsening of digital ulcers despite treatment | 24 months
  Healing: A novel composite outcome score for the assessment of worsening of digital ulcers despite treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marco Matucci-Cerinic, Prof., Principal Investigator — University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine; Francesco Del Galdo, Dr., Principal Investigator — The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital; Ulf Müller-Ladner, Prof., Study Chair — Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology
Locations (11):
- Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM 1016, Paris, France
- Germany (3):
  - Justus-Liebig-University Gießen, Kerckhoff Clinic, Departement of Rheumatology and Clinical Immunology, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Charité Centrum 12 für Innere Medizin und Dermatologie, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Centre for Pediatric Rheumatology, Klinikum Eilbek, Hamburg
- Pecsi Tudomanyegyetem - University of Pecs, Pécs, Hungary
- Italy (2):
  - University of Florence, Denothe Centre, Division of Rheumatology AOUC, Department of Biomedicine, Florence
  - Policlinico, Via Pansini, Napoli-Italia
- Switzerland (2):
  - Felix-Platter Spital, University of Basel, Basel
  - University of Zurich, Department of Rheumatology, Zurich
- United Kingdom (2):
  - The Universitiy of Leeds, Division of Rheumatic and Musculoskeletal Disease, St James's University Hospital, Leeds
  - Royal Free Hospital, University College London, London

REFERENCES:
- [Derived] Blagojevic J, Bellando-Randone S, Abignano G, Avouac J, Cometi L, Czirjak L, Denton CP, Distler O, Frerix M, Guiducci S, Huscher D, Jaeger VK, Lorand V, Maurer B, Nihtyanova S, Riemekasten G, Siegert E, Tarner IH, Vettori S, Walker UA, Allanore Y, Muller-Ladner U, Del Galdo F, Matucci-Cerinic M; EUSTAR co-workers. Classification, categorization and essential items for digital ulcer evaluation in systemic sclerosis: a DeSScipher/European Scleroderma Trials and Research group (EUSTAR) survey. Arthritis Res Ther. 2019 Jan 24;21(1):35. doi: 10.1186/s13075-019-1822-1. PMID 30678703